CLINICAL TRIAL: NCT04879810
Title: Pilot Clinical Trial Investigating the Ability of Plant Exosomes +/- Curcumin to Abrogate Symptoms of Inflammatory Bowel Disease (IBD)
Brief Title: Plant Exosomes +/- Curcumin to Abrogate Symptoms of Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Susan Galandiuk, Principal Investigator and Director, Division of Colorectal Surgery, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15.0872
Record Dates: First submitted 2018-06-06; First posted 2021-05-10 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Irritable Bowel Disease
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Sigmoidoscopy; Biopsy

STUDY DESIGN:
Intervention Model Description: three Arms: 1. Ginger exosomes;2. Curcumin; 3. Ginger exosomes plus curcumin, Each PO daily times 28 days. All subjects will receive active treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ginger exosomes (Active Comparator): Study mixture will be taken PO daily times 28 days Sigmoidoscopy and biopsy, blood work, quality of life questionnaire
  Interventions: Procedure: Sigmoidoscopy and biopsy, blood work
- Curcumin (Active Comparator): Study mixture will be taken PO daily times 28 days Sigmoidoscopy and biopsy, blood work, quality of life questionnaire
  Interventions: Procedure: Sigmoidoscopy and biopsy, blood work
- Ginger exosomes plus curcumin (Active Comparator): Study mixture will be taken PO daily times 28 days Sigmoidoscopy and biopsy, blood work, quality of life questionnaire
  Interventions: Procedure: Sigmoidoscopy and biopsy, blood work

INTERVENTIONS:
Procedure: Sigmoidoscopy and biopsy, blood work — Flexible tube up lower colon, blood draws, quality of life questionnaires
  Other Names: Inflammatory Bowel Disease Questionnaire

SUMMARY:
The trial will test the hypothesis that edible structures within plant cells (ginger) will have clinically important anti-inflammatory effects on the gut lining of patients with inflammable bowel disease.

To evaluate the safety and tolerability of exosomes with and without curcumin in patients with Inflammatory Bowel Disease (IBD); To estimate the effect of ginger exosomes or curcumin alone or combined with curcumin on the symptoms and disease score in patients with refractory IBD describe toxicities associated with ginger exosomes; to evaluate the effect of ginger exosomes on biomarkers of inflammation.

DETAILED DESCRIPTION:
Up to 90 patients with Chronic IBD will be enrolled, with the goal of having three arms of 30 subjects in each group who are eligible for evaluation.

This exploratory trial is designed to estimate the effect of ginger exosomes or curcumin on IBD symptoms compared to ginger exosomes plus curcumin. In this prospective and randomized study the main focus is to compare exosomes alone, curcumin, and exosomes plus curcumin. Three primary stratification factors race (white and black), gender and type of IBD (CD and UC) will be used. plan Zelen's (1974) method will be used to avoid imbalance allocation within each stratum. A block size of 4 will be used. We plan to enroll all eligible patients visiting the clinic, as well as eligible patients referred from other gastroenterologists. All eligible visiting our clinic will be enrolled. By enrolling consecutive patients, we reduce selection bias. A patient will be enrolled only once.

The most important aim of this study is to compare the IBD symptoms in exosomes alone and exosomes plus curcumin groups of patients. The symptomatology will be measured in each group and compared to the self-reported score. We will use the incidence rate of bloody stool to justify the sample size. With the combination treatment (ginger exosomes plus curcumin as compared to curcumin alone) we hope to reduce symptoms by at least 30%. Using a two sample one-sided t test for comparing mean differences in Inflammatory Bowel Disease Questionnaire, with 30 subjects in each group and using alpha=5%, we will have 80% power to detect effect size of 0.65 Standard Deviation, which is a large effect size (Cohen, 1988).. When the reduction in sample size due to missing data or other reasons, we will have reduced power to detect the difference in two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of IBD (either CD or UC) with moderate disease activity.)
* Ability to independently care for oneself

Exclusion Criteria:

* Pregnancy
* Known HIV
* Patients receiving immunosuppressive drugs, other than for their bowel disease
* Patients must be on stable doses of their medications for the 2 weeks prior to study entry and for the duration of the treatment period, or inform the investigator of any changes in medication
* Active malignancy in the last 5 years
* Patients receiving any other investigational agent(s)
* Ginger allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Change in inflammation on Colonoscopy | 30 days
  Decrease in inflammatory cells in the biopsy after treatment versus before treatment.

SECONDARY OUTCOMES:
Change in Subjective symptoms | 30 days
  Questionnaire reporting of decrease in subjective symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Galandiuk, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang M, Viennois E, Prasad M, Zhang Y, Wang L, Zhang Z, Han MK, Xiao B, Xu C, Srinivasan S, Merlin D. Edible ginger-derived nanoparticles: A novel therapeutic approach for the prevention and treatment of inflammatory bowel disease and colitis-associated cancer. Biomaterials. 2016 Sep;101:321-40. doi: 10.1016/j.biomaterials.2016.06.018. Epub 2016 Jun 9. PMID 27318094